CLINICAL TRIAL: NCT04223297
Title: Interest Assessment of the Blue Protocol in Improving Diagnosis of Dyspneic Patients in Pre- and Intra-hospital Emergency Medicine
Brief Title: Blue Protocol Assessment
Acronym: Blue P
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier de Clermont (Unknown); Centre Hospitalier de Montreuil sur Mer (Unknown); Centre Hospitalier de Beauvais (Other); Centre Hospitalier de Compiègne (Unknown); Centre Hospitalier de Doullens (Unknown); Centre Hospitalier de Abbeville (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0046
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Dyspnea; Emergencies
Keywords: dyspnea; lung ultrasound; emergency medicine; blue protocol
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lung ultrasound — The lung ultrasound will be performed by following the " Blue protocol "

SUMMARY:
Acute dyspnea is a common disease in emergency medicine. Mortality remains high is estimated at 15%. One third of initial diagnoses before paraclinical examination are estimated to be inaccurate. Lung ultrasound is a quick and immediate examination. Also, it is provided and performed at the bedside. The " Blue protocol " was designed by Daniel A. Lichtenstein as a diagnostic aid in dyspneic patients. It allows to obtain a diagnostic in more than 90% of acute dyspnea. However there is no validation in emergency medicine.

The main purpose is to evaluate the interest of the " Blue protocol "in the management and orientation of the dyspneic patient

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* dyspneic patient requiring management by an emergency physician
* information given and no patient opposition.

Exclusion Criteria:

* patient under a legal protection measure
* lack of social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each dyspneic patient meeting the inclusion criteria and admitted in emergency room will be included in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
concordance between the clinical diagnosis and the final diagnosis | day of arrival in emergency
  comparison of the concordance between the clinical diagnosis and the final diagnosis
concordance between the diagnosis establishes after the ultrasonography and the final diagnosis | day of arrival in emergency
  concordance between the diagnosis establishes after the ultrasonography and the final diagnosis

SECONDARY OUTCOMES:
Change of proportion of examinations leading to a change in the therapeutic hypothesis | 8 months
  Change of proportion of examinations leading to a change in the therapeutic hypothesis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No